CLINICAL TRIAL: NCT05876260
Title: Influence of Post-exercise Greek Yogurt on 24 h Glycemic Control in Women With Overweight/Obesity
Brief Title: Effect of Post-exercise Nutrition on Glycemia in Women
Acronym: PEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Jenna Gillen, Assistant Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 42756-3
Record Dates: First submitted 2023-05-05; First posted 2023-05-25 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Overweight and Obesity
Keywords: women; glycemic control; exercise
MeSH Terms: conditions — Overweight; Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval exercise and post-exercise Greek yogurt (HIIE+GY) (Experimental): Participants will consume greek yogurt following a single session of exercise
  Interventions: Behavioral: Greek yogurt; Behavioral: Exercise
- High-intensity interval exercise and post-exercise carbohydrate study supplement (HIIE +SS) (Active Comparator): Participants will consume a carbohydrate-based study supplement following a single session of exercise
  Interventions: Behavioral: Carbohydrate-based study supplement; Behavioral: Exercise

INTERVENTIONS:
Behavioral: Greek yogurt — Following 2 days of controlled diet, participants will consume greek yogurt following high-intensity interval exercise
  Arms: High-intensity interval exercise and post-exercise Greek yogurt (HIIE+GY)
Behavioral: Carbohydrate-based study supplement — Following 2 days of controlled diet, participants will consume a carbohydrate-based study supplement following high-intensity interval exercise
  Arms: High-intensity interval exercise and post-exercise carbohydrate study supplement (HIIE +SS)
Behavioral: Exercise — Following 2 days of controlled diet, participants will perform high-intensity interval exercise following an overnight fast

SUMMARY:
The purpose of this study is to assess whether post-exercise Greek yogurt following a single session of aerobic exercise improves metabolic and musculoskeletal health in women with overweight/obesity.

DETAILED DESCRIPTION:
Following the acquisition of informed consent, eligibility to participate in the study will be determined using questionnaires. Participants will undergo baseline testing at our laboratory at the University of Toronto to determine cardiorespiratory fitness, body composition and undergo exercise familiarization.

Eligible participants will be assigned, in a random order, to two metabolic trials approximately 4 weeks apart that involve 4 days of controlled diet and exercise. Each trial takes place over 4 days, but participants are not required to come to the laboratory on all days. The two trials involve: 1) Exercise + Greek Yogurt (GY) 2) Exercise + a carbohydrate-based study supplement (SS).

During the 4 day trials, participants consume controlled diets and the study supplements (GY and SS). On 1 of these days participants will perform exercise in our lab followed by the consumption of GY or SS. Various outcomes will be measured throughout the trial, including glycemic control (via continuous glucose monitoring), fat oxidation, appetite and health outcomes in blood samples.

Throughout the duration of the study, participants will be asked to maintain their habitual diet and physical activity patterns, and maintain their current body weight.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 yrs
* BMI ≥27 kg/m2
* Elevated waist circumference (≥88 cm)
* ≤2 structured exercise sessions/week
* Weight stable (within ± 2kg for at least 6 months)
* Experiencing regular natural menstrual cycles
* Non-smoker

Exclusion Criteria:

* Allergy to dairy foods
* Diagnosed lactose intolerance or an aversion to foods provided during the study (e.g., post-exercise snacks)
* Previous history of cardiovascular or metabolic disease
* The use of medication for managing blood glucose or lipid metabolism
* Current use of oral contraceptives or use within the last 3 months
* Irregular menstrual cycles (<21 days or >35 days)
* Pregnant or lactating
* Recreational tobacco or cannabis use
* Inability to perform the study exercise protocols
* Actively engaging in a low-carbohydrate diet (e.g., ketogenic, Atkins).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Postprandial glycemia | 24 hour post-exercise
  Postprandial glucose exposure assessed using continuous glucose monitoring

SECONDARY OUTCOMES:
24 hours average glucose | 24 hours post-exercise
  Average glucose concentration over 24 hours
Nocturnal glucose | 6-8 hours
  Overnight glucose concentration
Nocturnal glucose | 6-8 hours
  Overnight glucose exposure (area under the curve)
Glycemic variability | 24 hours
  Continuous overall net glycemic action (CONGA)
Glycemic variability | 24 hours
  Standard deviation (SD)
Glycemic variability | 24 hours
  Coefficient of variation (%CV)
Post-exercise fat oxidation | 1, 2 and 3 hours post-exercise
  Fat oxidation assessed with indirect calorimetry
Fasting glucose concentration | 24 hours post-exercise
  Venous blood sampling
Fasting insulin concentration | 24 hours post-exercise
  Venous blood sampling
Fasting insulin resistance | 24 hours post-exercise
  Homeostasis Model Assessment (HOMA2)
Bone metabolism | 30, 90, and 180 minutes and 24 hours post-exercise
  Serum concentration of CTX
Bone metabolism | 30, 90, and 180 minutes and 24 hours post-exercise
  Serum concentration of OPG
Bone metabolism | 30, 90, and 180 minutes and 24 hours post-exercise
  Serum concentration of RANKL
Bone metabolism | 30, 90, and 180 minutes and 24 hours post-exercise
  Serum concentration of OC

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Gillen, PhD, Principal Investigator — University of Toronto
Locations (1):
- Jenna Gillen, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No